CLINICAL TRIAL: NCT01479725
Title: A Prospective Trial Comparing the Response to Hyperbaric Oxygen Treatment in Patients With Ulcerative and Non-Ulcerative Interstitial Cystitis
Brief Title: Prospective Trial Comparing Response to Hyperbaric Oxygen Treatment in Patients With Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-247
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Interstitial Cystitis
Keywords: interstitial cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ulcerative IC (Experimental): HBOT for ulcerative IC
  Interventions: Procedure: HBOT
- Non-Ulcerative IC (Experimental): HBOT for non-ulcerative IC
  Interventions: Procedure: HBOT

INTERVENTIONS:
Procedure: HBOT — HBOT
  Other Names: hyperbaric oxygen therapy

SUMMARY:
To review the results of Hyperbaric Oxygen therapy (HBOT) on the symptoms of interstitial cystitis (IC). To determine if there is greater symptom improvement in the ulcerative vs the non-ulcerative patients with interstitial cystitis.

DETAILED DESCRIPTION:
There are multiple published studies outside of the United States on HBOT for treatment of interstitial cystitis. None of these studies compares ulcerative IC and non-ulcerative IC.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial cystitis.
* Urinary frequency of at least 8 times per 24 hours period.
* Patients with ulcerative IC must have undergone previous biopsy negative for cancer.
* Patients must agree to not begin any additional treatment for IC until study completion.

Exclusion Criteria:

* Absolute or relative contraindication to hyperbaric oxygen treatment.
* Patients dependent on intermittent catheterization or indwelling catheter to empty bladder.
* Any imminent change in residence, which could compromise compliance.
* Unlikely to be compliant due to unmanaged medical or psychological problems.
* Severe debilitating concurrent medical conditions.
* A history of pelvic radiation, bladder stone, bladder cancer or cancer in situ, or urethral cancer.
* Precious bladder or neurologic surgery which has affected bladder function.
* Currently has an active urethral stone, ureteral stone or urethral diverticulum.
* Subject misses more than 10 treatments.
* Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital, Royal Oak
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ulcerative IC | Non-Ulcerative IC
Started | 6 | 2
Completed | 4 | 1
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ulcerative IC | Non-Ulcerative IC | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [35 to 66] | 53 [51 to 55] | 54 [35 to 66]
Gender [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment (GRA)
Description: The GRA measures overall improvement with therapy. The patient's response describes their current condition compared to before they received hyperbaric oxygen therapy (HBOT). Responses are: 1 Markedly Worse, 2 Moderately Worse, 3 Mildly Worse, 4 Unchanged, 5 Mildly Better, 6 Moderately Better and 7 Markedly Better.
Time Frame: 3 months post treatment
Measure: Number; unit: number of participants
Arm/Group | Ulcerative IC | Non-Ulcerative IC
Number analyzed (Participants) | 6 | 2
number of participants
  Markedly Better | 0 | 1
  Moderately Better | 1 | 0
  Mildly Better | 4 | 0
  Unchanged | 0 | 1
  Mildy Worse | 0 | 0
  Moderately Worse | 0 | 0
  Markedly Worse | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ulcerative IC | Non-Ulcerative IC
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2

LIMITATIONS AND CAVEATS:
A small number of patients were enrolled and treated (n=8), with only 5 patients completing the entire study. Three patients withdrew within the year following HBOT and were considered non-responders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No